CLINICAL TRIAL: NCT04574583
Title: Phase I/II Trial Investigating the Safety, Tolerability, Pharmacokinetics, Immune and Clinical Activity of SX-682 in Combination With BinTrafusp Alfa (M7824 or TGF-beta "Trap"/PD-L1) With CV301 TRICOM in Advanced Solid Tumors (STAT)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, James Gulley, M.D., Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 200155; 20-C-0155
Record Dates: First submitted 2020-10-02; First posted 2020-10-05 (Actual); Results first posted 2023-05-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Cancer; Solid Tumors
Keywords: Immunotherapy; Checkpoint Inhibitor; Vaccine; Combination Therapy; Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis | interventions — bintrafusp alfa protein, human; smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase I Dose Level 1(DL1) 25mg SX-682 monotherapy sequentially foll/by 1200mg BinTraFusp Alfa +CV301 (Experimental): Participants with any solid tumor will receive a 2- week monotherapy lead-in of SX-682 DL2 50 mg by mouth (PO) twice a day (BID) followed sequentially by treatment with a dual combination of + BinTrafusp Alfa (M7824) 1200 mg fixed dose intravenous (IV) + BN-CV301.
  Participants will be evaluated for dose-limiting toxicities at the completion of the dose level before enrollment to the next dose level begins
  Interventions: Drug: SX-682; Drug: M7824; Biological: MVA-BN-CV301; Biological: recombinant fowlpox viral (FPV)-CV301
- Phase I Dose Level 2 (DL2) 50 mg SX-682 sequentially followed by 1200mg BinTraFusp Alfa + CV301 (Experimental): Participants with any solid tumor will receive a 2- week monotherapy lead-in of SX-682 DL2 50 mg by mouth (PO) twice a day (BID) followed sequentially by treatment with a dual combination of + BinTrafusp Alfa (M7824) 1200 mg fixed dose intravenous (IV) + BN-CV301.
  Participants will be evaluated for dose-limiting toxicities at the completion of the dose level before enrollment to the next dose level begins
  Interventions: Drug: SX-682; Drug: M7824; Biological: MVA-BN-CV301; Biological: recombinant fowlpox viral (FPV)-CV301
- Phase I Dose Level 3 (DL3) 100 mg SX-682 sequentially followed by 1200mg BinTraFusp Alfa +CV301 (Experimental): Participants with any solid tumor will receive a 2- week monotherapy lead-in of SX-682 DL1 100 mg by mouth (PO) twice a day (BID) followed sequentially by treatment with a dual combination of + BinTrafusp Alfa (M7824) 1200 mg fixed dose intravenous (IV) + BN-CV301.
  Participants will be evaluated for dose-limiting toxicities at the completion of the dose level before enrolling onto the next dose level.
  Interventions: Drug: SX-682; Drug: M7824; Biological: MVA-BN-CV301; Biological: recombinant fowlpox viral (FPV)-CV301

INTERVENTIONS:
Drug: SX-682 — SX-682 will be given orally at designated dose twice a day every day
Drug: M7824 — Subjects will receive M7824 at a flat dose of 1,200 mg intravenously on Days 1 and 15 of each cycle.
  Other Names: BinTrafusp Alfa
Biological: MVA-BN-CV301 — MVA-BN-CV301 will be given as four subcutaneous injections (4x10^8 Inf.U/0.5ml twice during Cycle 1 (Days 1 and 15)
  Other Names: modified vaccinia Ankara (MVA)-BN-CV301
Biological: recombinant fowlpox viral (FPV)-CV301 — FPV-CV301 will be given as one subcutaneous injection (1x10^9 Inf.U/0.5ml) on Day 1 starting at cycle 2 through cycle 5 (every 4 weeks) then on Day 1 of every 3 cycles (Cycles 8 and Cycle 11).

SUMMARY:
Background:

Combination immunotherapy techniques are being explored to improve responses and enhance benefits in people with cancer. Researchers want to see if this type of treatment can help people with advanced solid tumors.

Objective:

To find a safe dose of SX-682 in combined treatment with Bintrafusp alfa and BN-CV301 vaccines and to see if this treatment will cause tumors to shrink.

Eligibility:

Adults age 18 and older with metastatic cancer may be eligible for the first part of the trial. Adults age 18 and older with metastatic triple negative breast cancer or p16 negative head and neck squamous cell cancer, and who are not candidates for curative surgery may be eligible for the second part of the trial.

Design:

Participants will be screened under a separate protocol.

Participants may have tumor biopsies. They will have physical exams. Their symptoms and medicines will be reviewed. They will have blood tests. They will have electrocardiograms to evaluate their heart.

Participants will have imaging scans of the chest, abdomen, and pelvis. They may have a procedure where a small tube with a tiny video camera is put into the nose to look at the throat if they have head and neck cancers.

Participants will get bintrafusp alfa through an intravenous catheter. For this, a small tube is put into an arm vein. They will get BN-CV301 vaccines as injections in the arm or thigh. They will take SX-682 by mouth twice a day. They will take the study drugs up to 2 years. They will keep a medicine diary.

Participants will have study visits every 2 weeks. They will have 1 or 2 follow-up visits within 30 days after they stop treatment. Then they will be monitored by phone or email for 2 years.

DETAILED DESCRIPTION:
Background:

* Combination immunotherapy approaches are being actively explored to further improve responses, enhance clinical benefit, and overcome resistance to Programmed Cell Death Ligand 1 (PD(L)-1) agents in cancer participants.
* Interleukin-8 (IL-8) is a pro-inflammatory chemokine produced by various cell types. Overexpression of IL-8 and/or its receptors C-X-C motif chemokine receptor 1 (CXCR1) and C-X-C motif chemokine receptor 2 (CXCR2), is commonly seen in many human cancers including breast, cervical, melanoma and prostate.
* SX-682 is an oral, small molecule inhibitor of the CXCR1/2 chemokine receptors that are believed involved in myeloid-derived suppressor cells (MDSC)-recruitment to tumor and other pro-tumoral mechanisms.
* Bintrafusp alfa (M7824 or MSB0011359C) is a bifunctional protein composed of the extracellular domain of the Transforming Growth Factor Beta Receptor 2 (TGF-BetaRII) receptor (TGF-Beta 'trap') fused to a human immunoglobulin G1 (IgG1). Preclinical data shows bintrafusp alfa treatment increases T-cell trafficking, antigen specific cluster of differentiation 8 (CD8+) T-cell lysis and natural killer (NK) cell activation.
* CV301 is a poxviral-based vaccine comprised of recombinant Modified vaccinia Ankara (MVA-BN-CV301, prime) and recombinant fowlpox (FPV-CV301, boost). CV301 contains transgenes encoding two (2) tumor-associated antigens (TAA), mucin 1 (MUC1) and carcinoembryonic antigen (CEA), as well as three costimulatory molecules (B7.1, intercellular adhesion molecule 1 (ICAM-1) and lymphocyte function-associated antigen 3 (LFA-3), designated TRICOM). A recent phase 1 clinical trial demonstrated that antigen-specific T cells to MUC1 and CEA, as well as to a cascade antigen, brachyury, were generated in most participants.
* Preclinical studies performed in LTIB with SX-682, M7824 and a CEA-based vaccine showed a significant reduction in tumor growth as well as a significant increase in tumor infiltration with cluster of differentiation 4 (CD4+) and CD8+ T cells.

Objectives:

* Arm 1 (Sequential Dose Escalation):

  * To evaluate the safety and tolerability of single agent SX-682 given for 2 weeks preceding M7824 and CV301.
  * To determine the maximum tolerated dose (MTD) of SX-682 given for 2 weeks preceding M7824 and the CV301 vaccines in participants with advanced or metastatic solid tumors. If the MTD is not reached the study will be focused to describe the safety and tolerability of SX-682 followed by M7824 and CV301 vaccines.
* Arm 2 (Combination Dose Escalation):

  --To determine the recommended phase 2 dose (RP2D) of SX-682 given concurrently with M7824 and the CV301 vaccines in participants with advanced or metastatic solid tumors. If the MTD is not reached the study will be focused to describe the safety and tolerability of the drug combination.
* Arm 3 (Expansion):

  * To evaluate preliminary efficacy based on Objective Response Rate (ORR), in each disease separately in two cohorts: Triple Negative Breast Cancer (TNBC) and Human papilloma virus (HPV) negative head and neck squamous cell carcinoma (HNSCC).

Eligibility:

* Age >= 18 years old
* Arms 1 and 2 (Dose-Escalation Cohort): Subjects with cytologically or histologically confirmed locally advanced or metastatic solid tumors.
* Arm 3 (Expansion Cohorts):

  * Triple Negative Breast Cancer (TNBC): Subjects with cytologically or histologically confirmed locally advanced or metastatic Triple Negative Breast Cancer that has progressed on at least one prior treatment in the advanced or in the metastatic setting.
  * Human papilloma virus (HPV) negative head and neck squamous cell carcinoma (HNSCC): Subjects with cytologically or histologically confirmed locally advanced or metastatic, HPV negative head and neck squamous cell cancer (p16 negative for oropharyngeal) that has progressed on at least one prior treatment involving a platinum drug or cetuximab in advanced or in the metastatic setting.
* Prior first line systemic therapy is required unless there is no standard treatment available, the participant cannot tolerate standard first line treatment, or the participant declines standard treatment after appropriate counseling has been provided.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Adequate renal, hepatic, and hematologic function
* Subjects in Arms 1 and 2 may have disease that is measurable or non-measurable but evaluable disease (e.g. present on bone scan, rising tumor markers, non-measurable by Response Evaluation Criteria in Solid Tumors (RECIST) but visible on computed tomography (CT) scan). Participants with third space fluid (for example pleural effusions) as only site of disease will not be eligible. Subjects in Arm 3 must have measurable disease according to RECIST 1.1

Design:

* Arm 1 is a phase I, open-label, 3+3 sequential dose escalation trial with short term, 2-week SX-682 monotherapy, sequentially followed by treatment with M7824 and the CV301 vaccine series in advanced solid tumors (every 2 weeks (Q2W) dosing schedule) for the duration of treatment.
* Arm 2 is a phase I, open-label, 3+3 combination dose escalation trial with concurrently administered SX-682, M7824 and CV301 in advanced solid tumors (Q2W dosing schedule).
* Arm 3 has two expansion cohorts. Following identification of the MTD or recommended phase 2 dose (R2PD) for the combination of SX-682, M7824 and CV301 vaccine given concurrently, disease-specific phase 2 expansion cohorts will open in 1) advanced/metastatic triple negative breast cancer and 2) advanced/metastatic, platinum-refractory HPV negative head and neck squamous cell carcinoma.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must have histologically or cytologically confirmed:

  * Metastatic or locally advanced, Solid tumor (Cohort 1)

OR

--Metastatic or locally recurrent, non-resectable Triple Negative Breast Cancer (TNBC), defined as estrogen receptor (ER) < 10%, progesterone receptor (PR) < 10% per immunohistochemistry (IHC) and human epidermal growth factor receptor 2 (HER2) negative. HER2 negative or unamplified breast cancer is defined as IHC 0 or 1+ or IHC 2+ with FISH average HER2 copy number < 4.0 signals per cell or HER2/chromosome 17 (CEP17) < 2.0 with average HER2 copy number < 4.0 signals per cell.[89] HER2 testing must have been performed in a laboratory accredited by the College of American Pathology (CAP) or another accrediting entity (Cohort 2).

OR

* Metastatic or locally recurrent, non-resectable p16 negative Head and Neck Squamous Cell Cancer (HNSCC). Oropharyngeal tumors must be negative for p16 overexpression by IHC per American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines and in a CAP accredited lab.[90] All other head and neck malignancies do not require p16 testing (Cohort 3).

  * Participants must have histologically or cytologically confirmed metastatic or locally advanced disease. Historical reports from a CAP accredited lab are acceptable.
  * Subjects in Arms 1 and 2 may have disease that is measurable or non-measurable but evaluable disease (e.g. present on bone scan, rising tumor markers, non-measurable by Response Evaluation Criteria in Solid Tumors (RECIST) but visible on computed tomography (CT) scan). Participants with third space fluid (for example pleural effusions) as only site of disease will not be eligible. Subjects in Arm 3 must have measurable disease according to RECIST 1.1
  * Participants must
* have received at least one prior systemic therapy for metastatic or locally advanced disease, unless there is no standard treatment available,

OR

--not tolerate standard first line treatment,

OR

--decline standard treatment after appropriate counseling has been provided.

Note: Participants in Arm 3, Cohort 3 who have programmed death-ligand 1 (PD-L1) positive triple-negative breast cancer (TNBC) must have progressed on atezolizumab + nab-paclitaxel. Participants in Arm 3, Cohort 3 (p16 negative head and neck squamous cell carcinomas (HNSCC) must have progressed on or been intolerant to a regimen involving a platinum drug or cetuximab monotherapy.

* Age greater than or equal to 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Participants must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count (ANC) >1,500/mcL
  * Platelets >100,000/mcL
  * Hemoglobin > 9 g/dL without a blood transfusion in the 14 days prior to enrollment.
  * Total bilirubin < 1.5X upper limit of normal (ULN) OR in subjects with Gilbert s Syndrome, a total bilirubin < 3.0 x ULN
  * Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) serum glutamic-pyruvic aminotransaminase (SGPT) <2.5 X institutional upper limit of normal OR in subjects with known liver metastasis, AST/ALT < 3.0 X ULN
  * An estimated creatinine clearance (CrCl) > 60 mL/min/1.73 m^2 using the Cockcroft-Gault calculation (https://www.kidney.org/professionals/KDOQI/gfr_calculatorCoc).
* The effects of immunotherapies on the developing human fetus are unknown. For this reason and because immunotherapy agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) at the time of study entry, for the duration of study treatment and up to 6 months after the last dose of the study drug (s). Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Participants with well-controlled human immunodeficiency virus (HIV) infection are eligible for trial as long as:

  * On an effective anti-retroviral therapy (ART) > 4 weeks and with evidence of viral suppression defined as HIV viral load < 400 copies/mL at enrollment
  * CD4+ count > 200 cells/microL at enrollment
* No reported opportunistic infections within 6 months prior to enrollment except for the following which will be allowed:

  * Esophageal candidiasis treated within last 6 months or currently improving with antifungal treatment
  * Oral and/or genital herpes simplex virus (HSV) treated within last 6 months or currently improving with antiviral treatment
  * Mycobacterium avium infection in last 6 months or that has been treated for at least 1month.
* Immunomodulating drugs must be discontinued at least 1 weeks prior to enrollment for recent short course use (less than or equal to 14 days) or discontinued at least 4 weeks prior to enrollment for long term use (> 14 days).
* Participants must have a received their last treatment > 4 weeks or 5 half-lives of the last treatment drug, whichever is shorter before starting on trial.
* Participants with known history of hepatitis B (HBV) infection are eligible for trial as long as the HBV viral load is undetectable.
* Patients with known history of hepatitis C (HCV) infection must have been treated and cured (viral load is undetectable). For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable or unquantifiable HCV ribonucleic acid (RNA) 12 weeks or longer after definitive treatment completion.
* Subjects must be able to understand and be willing to sign a written informed consent document.

EXCLUSION CRITERIA:

* Participants who are receiving any other investigational agents.
* Participants with active brain metastases or central nervous system metastasis (less than 28 days out from definitive radiotherapy or surgery of brain metastasis) are excluded from this clinical trial. However, patients with treated brain metastasis are eligible if there is no magnetic resonance imaging (MRI) evidence of progression for 6 weeks after treatment is complete and the MRI within 28 days prior to enrollment. Participants requiring immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalent) for palliation are excluded. Patients with evidence of intratumoral or peritumoral brain metastasis hemorrhage on screening imaging are also excluded unless the hemorrhage of brain metastases is grade < 1 and has been stable on two consecutive imaging scans.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to any of study drugs
* Steroid use or active autoimmune disease that might deteriorate when receiving an immunostimulatory agent with the exception of:

  * Diabetes type I, eczema, vitiligo, alopecia, psoriasis, hypo- or hyperthyroid disease or other mild autoimmune disorder not requiring immunosuppressive treatment;
  * Participants requiring hormone replacement with corticosteroid are eligible if the steroids are administered only for the purpose of adrenal insufficiency and at doses of <10 mg of prednisone or equivalent per day;
  * Administration of steroids for other conditions through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) is acceptable;
  * Participants on physiologic doses of systemic intravenous or oral corticosteroid therapy (greater than or equal to the equivalent of prednisone 10 mg/day.
  * The use of corticosteroids as premedication for contrast-enhanced studies which is allowed prior to enrollment.
* Participants with a history of serious intercurrent chronic or acute illness, such as cardiac or pulmonary disease, hepatic disease, bleeding diathesis or recent (within 3 months) clinically significant bleeding events or other illness considered by the Investigator as high risk for investigational drug treatment.
* History of second malignancy within 3 years of enrollment except for the following: adequately treated localized skin cancer, ductal carcinoma in situ, cervical carcinoma in situ, superficial bladder cancer or other localized malignancy which has been adequately treated.
* Receipt of any organ transplantation requiring ongoing immunosuppression including allogenic stem-cell transplant.
* Participants with bone metastases who have initiated denosumab or a bisphosphonate therapy within 28 days prior to enrollment. Continuation of prior therapy is allowed.
* Participants who have a corrected QT interval by Fridericia (QTcf) interval > 475 msec or > 480 msec with a bundle branch block (BBB) on screening electrocardiogram.
* Participants with a personal or family history of long-QT syndrome or are on a concomitant drug that is known to cause significant QTc prolongation within 2 weeks or 5 half-lives (whichever is shorter) of enrollment
* Participants with heart failure (New York Heart Association [NYHA] class III or IV) or cerebrovascular accident within one year or acute myocardial infarction within one year.
* Participants unwilling to accept blood products or blood transfusions as medically indicated. As there is a risk of severe bleeding with M7824, participants must be willing to receive blood transfusions if medically necessary for their own safety
* Any other condition, which would, in the opinion of the Principal Investigator indicated the subject is a poor candidate for the clinical trial or would jeopardize the subject or the integrity of the data obtained.
* Pregnant women are excluded from this study because study drugs potential for teratogenic or abortifacient effects are unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with study drugs, breastfeeding should be discontinued if the mother is treated with study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James L Gulley, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-C-0155.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The trial never reached the point of enrolling to phase 2. It stopped early before maximum tolerated dose (MTD) was reached.
Groups:
- Phase I Dose Level 1(DL1) 25mg SX-682 Monotherapy Sequentially Foll/by 1200mg BinTraFusp Alfa +CV301: Participants with any solid tumor will receive a 2- week monotherapy lead-in of SX-682 DL2 25 mg by mouth (PO) twice a day (BID) followed sequentially by treatment with a dual combination of + BinTrafusp Alfa (M7824) 1200 mg fixed dose intravenous (IV) + BN-CV301.
  Participants will be evaluated for dose-limiting toxicities at the completion of the dose level before enrollment to the next dose level begins
Period: Overall Study
Arm/Group | Phase I Dose Level 1(DL1) 25mg SX-682 Monotherapy Sequentially Foll/by 1200mg BinTraFusp Alfa +CV301 | Phase I Dose Level 2 (DL2) 50 mg SX-682 Sequentially Followed by 1200mg BinTraFusp Alfa + CV301 | Phase I Dose Level 3 (DL3) 100 mg SX-682 Sequentially Followed by 1200mg BinTraFusp Alfa +CV301
Started | 3 | 6 | 3
Completed | 3 | 6 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Dose Level 1(DL1) 25mg SX-682 Monotherapy Sequentially Foll/by 1200mg BinTraFusp Alfa +CV301 | Phase I Dose Level 2 (DL2) 50 mg SX-682 Sequentially Followed by 1200mg BinTraFusp Alfa + CV301 | Phase I Dose Level 3 (DL3) 100 mg SX-682 Sequentially Followed by 1200mg BinTraFusp Alfa +CV301 | Total
Number analyzed (Participants) | 3 | 6 | 3 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 5 | 2 | 9
  >=65 years | 1 | 1 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.53 (5.23) | 59.38 (6.08) | 54 (13.29) | 58.58 (7.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 5
  Male | 2 | 4 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 5 | 3 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 5 | 2 | 9
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicities (DLT)
Description: A DLT is defined as any one of the following adverse events (AEs), as defined by Common Terminology Criteria for Adverse Events (CTCAE v5.0), that is possibly attributable to study drugs by the Investigator, that occur within 28 days after the start of study therapy: Any Grade 4 (life threatening) AEs, except for example, laboratory values that are determined to not be clinically significant or single laboratory valued that resolve to Grade ≤ 1 or baseline grade within 7 days with adequate medical management. Average corrected QT interval by Fridericia (QTcF)≥ 501 msec or > 60 msec change from baseline (Grade 3). Any Grade 3 (severe) AEs except for example, Grade 3 flu-like symptoms or fever, as well as associated symptoms of fatigue, headaches, nausea, emesis which can be controlled with conservative medical management. Any grade 3 or higher adverse event or unexpected toxicities due to the combination of therapies that would not be expected with individual agents alone.
Time Frame: DLT observation period (first 4 weeks)
Measure: Number; unit: toxicities
Arm/Group | Phase I Dose Level 1(DL1) 25mg SX-682 Monotherapy Sequentially Foll/by 1200mg BinTraFusp Alfa +CV301 | Phase I Dose Level 2 (DL2) 50 mg SX-682 Sequentially Followed by 1200mg BinTraFusp Alfa + CV301 | Phase I Dose Level 3 (DL3) 100 mg SX-682 Sequentially Followed by 1200mg BinTraFusp Alfa +CV301
Number analyzed (Participants) | 3 | 6 | 3
toxicities | 0 | 1 | 0

2. Primary Outcome: Number of Participants With Grades 3-5 Adverse Events (AEs) Related and/or Unrelated to SX-682 + BinTrafusp Alfa (M7824) + BN-CV301
Description: Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). Grade 1 is mild. Grade 2 is moderate. Grade 3 is severe. Grade 4 is life-threatening. Grade 5 is death related to AE.
Time Frame: Approximately 16 months and 11 days
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level 1(DL1) 25mg SX-682 Monotherapy Sequentially Foll/by 1200mg BinTraFusp Alfa +CV301 | Phase I Dose Level 2 (DL2) 50 mg SX-682 Sequentially Followed by 1200mg BinTraFusp Alfa + CV301 | Phase I Dose Level 3 (DL3) 100 mg SX-682 Sequentially Followed by 1200mg BinTraFusp Alfa +CV301
Number analyzed (Participants) | 3 | 6 | 3
Participants
  Grade 3 Related | 2 | 2 | 2
  Grade 4 Related | 0 | 0 | 0
  Grade 5 Related | 0 | 0 | 0
  Grade 3 Unrelated | 1 | 4 | 2
  Grade 4 Unrelated | 0 | 0 | 0
  Grade 5 Unrelated | 0 | 1 | 0

3. Primary Outcome: Maximum Tolerated Dose (MTD) of SX-682 Followed by BinTrafusp Alfa (M7824) and CV301 Vaccines in Participants With Advanced or Metastatic Solid Tumors.
Description: The MTD is the dose at which no more than 1 of 6 subjects taking SX-682 followed by M7824 and CV301 vaccines experience a dose-limiting toxicity (DLT). A DLT is defined as any one of the following adverse events (AEs), as defined by Common Terminology Criteria for Adverse Events (CTCAE v5.0), that is possibly attributable to study drugs by the Investigator, that occur within 28 days after the start of study therapy.
Time Frame: Period of Safety lead-in (monotherapy), approximately 28 days
Measure: Number; unit: mg
Groups:
- All Participants: All participants with any solid tumor (e.g., triple negative breast cancer, and human papilloma virus (HPV) head and neck cancer) who received a 2-week monotherapy lead-in dose of 25mg, 50mg, and 100mg SX-682 by mouth (PO) twice a day (BID) followed by treatment with a dual combination of + BinTrafusp Alfa (M7824) + BN-CV301 respectively, were evaluated for dose-limiting toxicities at the completion of the dose level before enrolling onto the next dose level in an effort to determine the recommended phase 2 dose.
Arm/Group | All Participants
Number analyzed (Participants) | 12
mg | NA — The MTD was not established because the study was stopped due to toxicity.

4. Primary Outcome: Recommended Phase II Dose (RP2D) of SX-682 With BinTrafusp Alfa (M7824) and CV301 Vaccines in Participants With Advanced or Metastatic Solid Tumors.
Description: Recommended phase II dose is defined as the dose defined in the phase I portion of a study that will be administered to participants on the phase II portion.
Time Frame: Approximately 28 days
Measure: Number; unit: mg
Arm/Group | All Participants
Number analyzed (Participants) | 12
mg | NA — The RP2D was not established because the study was stopped due to toxicity.

5. Primary Outcome: Percentage of Participants Who Experience a Response
Description: The percentage of participants who experience a response will be reported along with 95% two-sided confidence intervals. The objective response is the best overall response recorded from the start of treatment until disease progression/recurrence per the Response Evaluation Criteria in Solid Tumors (RECIST). Complete Response is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Stable Disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study. Progressive Disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study.
Time Frame: 11 months
Population: 2 participants were not evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Groups:
- Phase I Solid Tumor Dose Level 1 (DL1) Sequential Dose Escalation: SX-682 DL1 25 mg by mouth (PO) twice a day (BID) + BinTrafusp Alfa (M7824) 1200 mg intravenous (IV) every 2 weeks (Q2 wk) + BN-CV301 Sequential Dose Escalation: Escalating doses of SX-682 for 2 weeks THEN M7824 + CV301
- Phase I Solid Tumor Dose Level 2 (DL2) Combination Dose Escalation: SX-682 DL1 50 mg by mouth (PO) twice a day (BID) + BinTrafusp Alfa (M7824) 1200 mg intravenous (IV) every 2 weeks (Q2 wk) + BN-CV301 Combination Dose Escalation: Escalating doses of SX-682 for 2 weeks THEN escalating doses of SX-682 + M7824 +CV301
- Phase I Solid Tumor Dose Level 3 (DL3) Disease-Specific Expansion: SX-682 DL1 100 mg by mouth (PO) twice a day (BID) + BinTrafusp Alfa (M7824) 1200 mg intravenous (IV) every 2 weeks (Q2 wk) + BN-CV301 Disease-Specific Expansion: Recommended phase 2 dose (RP2D) of SX-682+ M7824 + CV301
Arm/Group | Phase I Solid Tumor Dose Level 1 (DL1) Sequential Dose Escalation | Phase I Solid Tumor Dose Level 2 (DL2) Combination Dose Escalation | Phase I Solid Tumor Dose Level 3 (DL3) Disease-Specific Expansion
Number analyzed (Participants) | 3 | 5 | 2
percentage of participants
  Complete Response | 0 | 0 | 0
  Partial Response | 0 | 0 | 0
  Stable Disease | 100 | 60 | 0
  Progressive Disease | 100 | 40 | 100

6. Secondary Outcome: Percentage of Participants Disease Control Rate (DCR): Complete Response (CR)+ Partial Response (PR) + Stable Disease (SD)
Description: The percentage of participants disease control rate (DCR): Complete response (CR)+ partial response (PR) + stable disease (SD) was measured by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete Response is disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Stable Disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study. Progressive Disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: Date first participant enrolled and ending on the off treatment date of the last participant on treatment (i.e., assessed beyond the primary completion date), approximately 15 months and 14 days.
Population: 2 participants were not evaluable for this outcome measure. The Rows were not planned to be mutually exhaustive and consisted of only those participants with response.
Measure: Number; unit: percentage of participants
Arm/Group | Phase I Dose Level 1(DL1) 25mg SX-682 Monotherapy Sequentially Foll/by 1200mg BinTraFusp Alfa +CV301 | Phase I Dose Level 2 (DL2) 50 mg SX-682 Sequentially Followed by 1200mg BinTraFusp Alfa + CV301 | Phase I Dose Level 3 (DL3) 100 mg SX-682 Sequentially Followed by 1200mg BinTraFusp Alfa +CV301
Number analyzed (Participants) | 3 | 5 | 2
percentage of participants
  Complete Response | 0 | 0 | 0
  Partial Response | 0 | 0 | 0
  Stable Disease | 100 | 60 | 0

7. Secondary Outcome: Progression-free Survival (PFS) Using Response Evaluation Criteria in Solid Tumors (RECIST)1.1.
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Progression per the RECIST is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The appearance of one or more new lesions is also considered progressions.
Time Frame: Time from start of treatment to time of progression or death, whichever occurs first, approximately 10 months
Measure: Median (Full Range); unit: months
Arm/Group | Phase I Dose Level 1(DL1) 25mg SX-682 Monotherapy Sequentially Foll/by 1200mg BinTraFusp Alfa +CV301 | Phase I Dose Level 2 (DL2) 50 mg SX-682 Sequentially Followed by 1200mg BinTraFusp Alfa + CV301 | Phase I Dose Level 3 (DL3) 100 mg SX-682 Sequentially Followed by 1200mg BinTraFusp Alfa +CV301
Number analyzed (Participants) | 3 | 6 | 3
months | 2.0 [1.5 to 6.9] | 3.4 [1.0 to 10.4] | 1.8 [1.3 to 2.3]

8. Secondary Outcome: Pharmacokinetic Profile of SX-682 as a Single Agent and in Combination
Description: Plasma and serum samples will be drawn and may be analyzed by a validated immunoassay to quantitate SX-682 as a single agent and in combination or by a validated electrochemiluminescence immunoassay to detect the presence of M7824 concentration.
Time Frame: Predose, 30 minutes, 60 minutes, 120 minutes, <6 hours of 2nd dose, and end of infusion (EOI)
Population: Blood samples were collected on only a subset of participants because the study was closed to enrollment early due to a safety stopping rule pre-specified in the protocol. Since no participants received SX-682 treatment in combination, with bintrasfusp alfa and CV-301, the PK analysis cannot be performed completely as outlined in the study objectives. Below are analyses of all available participant samples.
Measure: Number; unit: ng/ml
Arm/Group | Phase I Dose Level 1(DL1) 25mg SX-682 Monotherapy Sequentially Foll/by 1200mg BinTraFusp Alfa +CV301 | Phase I Dose Level 2 (DL2) 50 mg SX-682 Sequentially Followed by 1200mg BinTraFusp Alfa + CV301 | Phase I Dose Level 3 (DL3) 100 mg SX-682 Sequentially Followed by 1200mg BinTraFusp Alfa +CV301
Number analyzed (Participants) | 3 | 6 | 3
ng/ml
  Participant 1 - PRE, Day 14: number analyzed (Participants) | 1 | 0 | 0
  Participant 1 - PRE, Day 14 | NA — Below quantifiable limit (BQL) |  |
  Participant 1 - 30 minutes, Day 14: number analyzed (Participants) | 1 | 0 | 0
  Participant 1 - 30 minutes, Day 14 | 7.88 |  |
  Participant 1 - 60 minutes, Day 14: number analyzed (Participants) | 1 | 0 | 0
  Participant 1 - 60 minutes, Day 14 | 17.7 |  |
  Participant 1 - 120 minutes, Day 14: number analyzed (Participants) | 1 | 0 | 0
  Participant 1 - 120 minutes, Day 14 | 104 |  |
  Participant 1 - 180 minutes, Day 14: number analyzed (Participants) | 1 | 0 | 0
  Participant 1 - 180 minutes, Day 14 | 124 |  |
  Participant 1 - <6 hours (HR) of 2nd dose, Day 14: number analyzed (Participants) | 1 | 0 | 0
  Participant 1 - <6 hours (HR) of 2nd dose, Day 14 | 105 |  |
  Participant 1 - PRE, Day 7: number analyzed (Participants) | 1 | 0 | 0
  Participant 1 - PRE, Day 7 | 214 |  |
  Participant 1 - 30 minutes, Day 7: number analyzed (Participants) | 1 | 0 | 0
  Participant 1 - 30 minutes, Day 7 | 193 |  |
  Participant 1 - PRE, Cycle 1 Day 1 (C1D1): number analyzed (Participants) | 1 | 0 | 0
  Participant 1 - PRE, Cycle 1 Day 1 (C1D1) | 325 |  |
  Participant 1 - End of infusion (EOI), C1D1: number analyzed (Participants) | 1 | 0 | 0
  Participant 1 - End of infusion (EOI), C1D1 | 116 |  |
  Participant 1 - PRE, Cycle 1 Day 15 (C1D15): number analyzed (Participants) | 1 | 0 | 0
  Participant 1 - PRE, Cycle 1 Day 15 (C1D15) | NA — Below quantifiable limit (BQL) |  |
  Participant 1 - PRE, Cycle 2 Day 1 (C2D1): number analyzed (Participants) | 1 | 0 | 0
  Participant 1 - PRE, Cycle 2 Day 1 (C2D1) | NA — Below quantifiable limit (BQL) |  |
  Participant 2 - PRE, Day 14: number analyzed (Participants) | 1 | 0 | 0
  Participant 2 - PRE, Day 14 | NA — Below quantifiable limit (BQL) |  |
  Participant 2 - 30 minutes, Day 14: number analyzed (Participants) | 1 | 0 | 0
  Participant 2 - 30 minutes, Day 14 | 216 |  |
  Participant 2 - 60 minutes, Day 14: number analyzed (Participants) | 1 | 0 | 0
  Participant 2 - 60 minutes, Day 14 | 460 |  |
  Participant 2 - 120 minutes, Day 14: number analyzed (Participants) | 1 | 0 | 0
  Participant 2 - 120 minutes, Day 14 | 483 |  |
  Participant 2 - 180 minutes, Day 14: number analyzed (Participants) | 1 | 0 | 0
  Participant 2 - 180 minutes, Day 14 | 448 |  |
  Participant 2 - <6 hours (HR) of 2nd dose, Day 14: number analyzed (Participants) | 1 | 0 | 0
  Participant 2 - <6 hours (HR) of 2nd dose, Day 14 | 184 |  |
  Participant 2 - PRE, Day 7: number analyzed (Participants) | 1 | 0 | 0
  Participant 2 - PRE, Day 7 | 421 |  |
  Participant 2 - 30 minutes, Day 7: number analyzed (Participants) | 1 | 0 | 0
  Participant 2 - 30 minutes, Day 7 | 394 |  |
  Participant 2 - PRE, Cycle 1 Day 1 (C1D1): number analyzed (Participants) | 1 | 0 | 0
  Participant 2 - PRE, Cycle 1 Day 1 (C1D1) | 778 |  |
  Participant 2 - End of infusion (EOI), C1D1: number analyzed (Participants) | 1 | 0 | 0
  Participant 2 - End of infusion (EOI), C1D1 | 587 |  |
  Participant 2 - PRE, Cycle 1 Day 15 (C1D15): number analyzed (Participants) | 1 | 0 | 0
  Participant 2 - PRE, Cycle 1 Day 15 (C1D15) | 1.24 |  |
  Participant 3 - PRE, Day 14: number analyzed (Participants) | 1 | 0 | 0
  Participant 3 - PRE, Day 14 | NA — Below quantifiable limit (BQL) |  |
  Participant 3 - 30 minutes, Day 14: number analyzed (Participants) | 1 | 0 | 0
  Participant 3 - 30 minutes, Day 14 | NA — Below quantifiable limit (BQL) |  |
  Participant 3 - 60 minutes, Day 14: number analyzed (Participants) | 1 | 0 | 0
  Participant 3 - 60 minutes, Day 14 | 6.13 |  |
  Participant 3 - 120 minutes, Day 14: number analyzed (Participants) | 1 | 0 | 0
  Participant 3 - 120 minutes, Day 14 | 31.3 |  |
  Participant 3 - 180 minutes, Day 14: number analyzed (Participants) | 1 | 0 | 0
  Participant 3 - 180 minutes, Day 14 | 65.6 |  |
  Participant 3- <6 hours (HR) of 2nd dose, Day 14: number analyzed (Participants) | 1 | 0 | 0
  Participant 3- <6 hours (HR) of 2nd dose, Day 14 | 99.7 |  |
  Participant 3 - PRE, Day 7: number analyzed (Participants) | 1 | 0 | 0
  Participant 3 - PRE, Day 7 | 53.7 |  |
  Participant 3 - 30 minutes, Day 7: number analyzed (Participants) | 1 | 0 | 0
  Participant 3 - 30 minutes, Day 7 | 51.2 |  |
  Participant 3 - PRE, Cycle 1 Day 1 (C1D1): number analyzed (Participants) | 1 | 0 | 0
  Participant 3 - PRE, Cycle 1 Day 1 (C1D1) | 170 |  |
  Participant 3 - End of infusion (EOI), C1D1: number analyzed (Participants) | 1 | 0 | 0
  Participant 3 - End of infusion (EOI), C1D1 | 84 |  |
  Participant 3 - PRE, Cycle 1 Day 15 (C1D15): number analyzed (Participants) | 1 | 0 | 0
  Participant 3 - PRE, Cycle 1 Day 15 (C1D15) | NA — Below quantifiable limit (BQL) |  |
  Participant 3 - PRE, Cycle 2 Day 1 (C2D1): number analyzed (Participants) | 1 | 0 | 0
  Participant 3 - PRE, Cycle 2 Day 1 (C2D1) | NA — Below quantifiable limit (BQL) |  |
  Participant 3 - PRE, Cycle 3 Day 1 (C3D1): number analyzed (Participants) | 1 | 0 | 0
  Participant 3 - PRE, Cycle 3 Day 1 (C3D1) | NA — Below quantifiable limit (BQL) |  |
  Participant 4 - PRE, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 4 - PRE, Day 14 |  | NA — Below quantifiable limit (BQL) |
  Participant 4 - 30 minutes, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 4 - 30 minutes, Day 14 |  | 10.9 |
  Participant 4 - 60 minutes, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 4 - 60 minutes, Day 14 |  | 38.2 |
  Participant 4 - 120 minutes, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 4 - 120 minutes, Day 14 |  | 148 |
  Participant 4 - 180 minutes, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 4 - 180 minutes, Day 14 |  | 160 |
  Participant 4 - <6 hours (HR) of 2nd dose, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 4 - <6 hours (HR) of 2nd dose, Day 14 |  | 225 |
  Participant 4 - PRE, Day 7: number analyzed (Participants) | 0 | 1 | 0
  Participant 4 - PRE, Day 7 |  | 710 |
  Participant 4 - 30 minutes, Day 7: number analyzed (Participants) | 0 | 1 | 0
  Participant 4 - 30 minutes, Day 7 |  | 827 |
  Participant 4 - PRE, Cycle 1 Day 1 (C1D1): number analyzed (Participants) | 0 | 1 | 0
  Participant 4 - PRE, Cycle 1 Day 1 (C1D1) |  | 902 |
  Participant 4 - End of infusion (EOI), C1D1: number analyzed (Participants) | 0 | 1 | 0
  Participant 4 - End of infusion (EOI), C1D1 |  | 501 |
  Participant 4 - PRE, Cycle 1 Day 15 (C1D15): number analyzed (Participants) | 0 | 1 | 0
  Participant 4 - PRE, Cycle 1 Day 15 (C1D15) |  | 1.56 |
  Participant 4 - End of treatment (EOT), Cycle 2 Day 1 (C2D1): number analyzed (Participants) | 0 | 1 | 0
  Participant 4 - End of treatment (EOT), Cycle 2 Day 1 (C2D1) |  | NA — Below quantifiable limit (BQL) |
  Participant 5 - PRE, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 5 - PRE, Day 14 |  | NA — Below quantifiable limit (BQL) |
  Participant 5 - 30 minutes, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 5 - 30 minutes, Day 14 |  | 11.9 |
  Participant 5 - 60 minutes, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 5 - 60 minutes, Day 14 |  | 27.4 |
  Participant 5 - 120 minutes, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 5 - 120 minutes, Day 14 |  | 439 |
  Participant 5 - 180 minutes, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 5 - 180 minutes, Day 14 |  | 706 |
  Participant 5 - <6 hours (HR) of 2nd dose, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 5 - <6 hours (HR) of 2nd dose, Day 14 |  | 419 |
  Participant 5 - PRE, Day 7: number analyzed (Participants) | 0 | 1 | 0
  Participant 5 - PRE, Day 7 |  | 1660 |
  Participant 5 - 30 minutes, Day 7: number analyzed (Participants) | 0 | 1 | 0
  Participant 5 - 30 minutes, Day 7 |  | 1940 |
  Participant 5 - PRE, Cycle 1 Day 1 (C1D1): number analyzed (Participants) | 0 | 1 | 0
  Participant 5 - PRE, Cycle 1 Day 1 (C1D1) |  | 3170 |
  Participant 5 - End of infusion (EOI), C1D1: number analyzed (Participants) | 0 | 1 | 0
  Participant 5 - End of infusion (EOI), C1D1 |  | 1660 |
  Participant 6 - PRE, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 6 - PRE, Day 14 |  | NA — Below quantifiable limit (BQL) |
  Participant 6 - 30 minutes, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 6 - 30 minutes, Day 14 |  | 32 |
  Participant 6 - 60 minutes, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 6 - 60 minutes, Day 14 |  | 219 |
  Participant 6 - 120 minutes, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 6 - 120 minutes, Day 14 |  | 395 |
  Participant 6 - 180 minutes, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 6 - 180 minutes, Day 14 |  | 341 |
  Participant 6 - <6 hours (HR) of 2nd dose, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 6 - <6 hours (HR) of 2nd dose, Day 14 |  | 260 |
  Participant 6 - PRE, Day 7: number analyzed (Participants) | 0 | 1 | 0
  Participant 6 - PRE, Day 7 |  | 679 |
  Participant 6 - 30 minutes, Day 7: number analyzed (Participants) | 0 | 1 | 0
  Participant 6 - 30 minutes, Day 7 |  | 777 |
  Participant 6 - PRE, Cycle 1 Day 1 (C1D1): number analyzed (Participants) | 0 | 1 | 0
  Participant 6 - PRE, Cycle 1 Day 1 (C1D1) |  | 683 |
  Participant 6 - End of infusion (EOI), C1D1: number analyzed (Participants) | 0 | 1 | 0
  Participant 6 - End of infusion (EOI), C1D1 |  | 429 |
  Participant 6 - PRE, Cycle 1 Day 15 (C1D15): number analyzed (Participants) | 0 | 1 | 0
  Participant 6 - PRE, Cycle 1 Day 15 (C1D15) |  | 1.25 |
  Participant 6 - PRE, Cycle 2 Day 1 (C2D1): number analyzed (Participants) | 0 | 1 | 0
  Participant 6 - PRE, Cycle 2 Day 1 (C2D1) |  | NA — Below quantifiable limit (BQL) |
  Participant 6 - PRE, Cycle 3 Day 1 (C3D1): number analyzed (Participants) | 0 | 1 | 0
  Participant 6 - PRE, Cycle 3 Day 1 (C3D1) |  | NA — Below quantifiable limit (BQL) |
  Participant 7 - PRE, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 7 - PRE, Day 14 |  | NA — Below quantifiable limit (BQL) |
  Participant 7 - 30 minutes, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 7 - 30 minutes, Day 14 |  | 97.1 |
  Participant 7 - 60 minutes, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 7 - 60 minutes, Day 14 |  | 110 |
  Participant 7 - 120 minutes, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 7 - 120 minutes, Day 14 |  | 54.2 |
  Participant 7 - 180 minutes, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 7 - 180 minutes, Day 14 |  | 705 |
  Participant 7 - <6 hours (HR) of 2nd dose, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 7 - <6 hours (HR) of 2nd dose, Day 14 |  | 489 |
  Participant 7 - PRE, Day 7: number analyzed (Participants) | 0 | 1 | 0
  Participant 7 - PRE, Day 7 |  | 1900 |
  Participant 7 - 30 minutes, Day 7: number analyzed (Participants) | 0 | 1 | 0
  Participant 7 - 30 minutes, Day 7 |  | 1870 |
  Participant 7 - PRE, Cycle 1 Day 1 (C1D1): number analyzed (Participants) | 0 | 1 | 0
  Participant 7 - PRE, Cycle 1 Day 1 (C1D1) |  | 1840 |
  Participant 7 - End of infusion (EOI), C1D1: number analyzed (Participants) | 0 | 1 | 0
  Participant 7 - End of infusion (EOI), C1D1 |  | 1070 |
  Participant 8 - PRE, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 8 - PRE, Day 14 |  | NA — Below quantifiable limit (BQL) |
  Participant 8 - 30 minutes, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 8 - 30 minutes, Day 14 |  | 8.68 |
  Participant 8 - 60 minutes, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 8 - 60 minutes, Day 14 |  | 394 |
  Participant 8 - 120 minutes, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 8 - 120 minutes, Day 14 |  | 467 |
  Participant 8 - 180 minutes, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 8 - 180 minutes, Day 14 |  | 443 |
  Participant 8 - <6 hours (HR) of 2nd dose, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 8 - <6 hours (HR) of 2nd dose, Day 14 |  | 199 |
  Participant 8 - PRE, Day 7: number analyzed (Participants) | 0 | 1 | 0
  Participant 8 - PRE, Day 7 |  | 480 |
  Participant 8 - 30 minutes, Day 7: number analyzed (Participants) | 0 | 1 | 0
  Participant 8 - 30 minutes, Day 7 |  | 455 |
  Participant 8 - PRE, Cycle 1 Day 1 (C1D1): number analyzed (Participants) | 0 | 1 | 0
  Participant 8 - PRE, Cycle 1 Day 1 (C1D1) |  | 465 |
  Participant 8 - End of infusion (EOI), C1D1: number analyzed (Participants) | 0 | 1 | 0
  Participant 8 - End of infusion (EOI), C1D1 |  | 478 |
  Participant 8 - PRE, Cycle 1 Day 15 (C1D15): number analyzed (Participants) | 0 | 1 | 0
  Participant 8 - PRE, Cycle 1 Day 15 (C1D15) |  | 1.54 |
  Participant 8 - PRE, Cycle 2 Day 1 (C2D1): number analyzed (Participants) | 0 | 1 | 0
  Participant 8 - PRE, Cycle 2 Day 1 (C2D1) |  | NA — Below quantifiable limit (BQL) |
  Participant 8 - PRE, Cycle 3 Day 1 (C3D1): number analyzed (Participants) | 0 | 1 | 0
  Participant 8 - PRE, Cycle 3 Day 1 (C3D1) |  | NA — Below quantifiable limit (BQL) |
  Participant 9 - PRE, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 9 - PRE, Day 14 |  | NA — Below quantifiable limit (BQL) |
  Participant 9 - 30 minutes, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 9 - 30 minutes, Day 14 |  | 2.63 |
  Participant 9 - 60 minutes, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 9 - 60 minutes, Day 14 |  | 37.9 |
  Participant 9 - 120 minutes, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 9 - 120 minutes, Day 14 |  | 113 |
  Participant 9 - 180 minutes, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 9 - 180 minutes, Day 14 |  | 305 |
  Participant 9 - <6 hours (HR) of 2nd dose, Day 14: number analyzed (Participants) | 0 | 1 | 0
  Participant 9 - <6 hours (HR) of 2nd dose, Day 14 |  | 350 |
  Participant 9 - PRE, Cycle 1 Day 1 (C1D1): number analyzed (Participants) | 0 | 1 | 0
  Participant 9 - PRE, Cycle 1 Day 1 (C1D1) |  | 424 |
  Participant 9 - End of infusion (EOI), C1D1: number analyzed (Participants) | 0 | 1 | 0
  Participant 9 - End of infusion (EOI), C1D1 |  | 416 |
  Participant 9 - PRE, Cycle 1 Day 15 (C1D15): number analyzed (Participants) | 0 | 1 | 0
  Participant 9 - PRE, Cycle 1 Day 15 (C1D15) |  | NA — Below quantifiable limit (BQL) |
  Participant 9 - PRE, Cycle 2 Day 1 (C2D1): number analyzed (Participants) | 0 | 1 | 0
  Participant 9 - PRE, Cycle 2 Day 1 (C2D1) |  | NA — Below quantifiable limit (BQL) |
  Participant 9 - Cycle 3 Day 1 (C3D1): number analyzed (Participants) | 0 | 1 | 0
  Participant 9 - Cycle 3 Day 1 (C3D1) |  | NA — Below quantifiable limit (BQL)/Treatment (tx) held |
  Participant 9 - PRE, Cycle 3 Day 1 (C3D1): number analyzed (Participants) | 0 | 1 | 0
  Participant 9 - PRE, Cycle 3 Day 1 (C3D1) |  | NA — Below quantifiable limit (BQL)/Treatment (tx) restart |
  Participant 10 - PRE, Day 14: number analyzed (Participants) | 0 | 0 | 1
  Participant 10 - PRE, Day 14 |  |  | NA — Below quantifiable limit (BQL)
  Participant 10 - 30 minutes, Day 14: number analyzed (Participants) | 0 | 0 | 1
  Participant 10 - 30 minutes, Day 14 |  |  | NA — Below quantifiable limit (BQL)
  Participant 10 - 60 minutes, Day 14: number analyzed (Participants) | 0 | 0 | 1
  Participant 10 - 60 minutes, Day 14 |  |  | 1.28
  Participant 10 - 120 minutes, Day 14: number analyzed (Participants) | 0 | 0 | 1
  Participant 10 - 120 minutes, Day 14 |  |  | 39.2
  Participant 10 - 180 minutes, Day 14: number analyzed (Participants) | 0 | 0 | 1
  Participant 10 - 180 minutes, Day 14 |  |  | 155
  Participant 10 - <6 hours (HR) of 2nd dose, Day 14: number analyzed (Participants) | 0 | 0 | 1
  Participant 10 - <6 hours (HR) of 2nd dose, Day 14 |  |  | 329
  Participant 10 - PRE, Day 7: number analyzed (Participants) | 0 | 0 | 1
  Participant 10 - PRE, Day 7 |  |  | 991
  Participant 10 - 30 minutes, Day 7: number analyzed (Participants) | 0 | 0 | 1
  Participant 10 - 30 minutes, Day 7 |  |  | 1220
  Participant 10 - PRE, Cycle 1 Day 1 (C1D1): number analyzed (Participants) | 0 | 0 | 1
  Participant 10 - PRE, Cycle 1 Day 1 (C1D1) |  |  | 923
  Participant 10 - End of infusion (EOI), C1D1: number analyzed (Participants) | 0 | 0 | 1
  Participant 10 - End of infusion (EOI), C1D1 |  |  | 745
  Participant 10 - PRE, Cycle 1 Day 15 (C1D15): number analyzed (Participants) | 0 | 0 | 1
  Participant 10 - PRE, Cycle 1 Day 15 (C1D15) |  |  | NA — Below quantifiable limit (BQL)
  Participant 11 - PRE, Day 14: number analyzed (Participants) | 0 | 0 | 1
  Participant 11 - PRE, Day 14 |  |  | NA — Below quantifiable limit (BQL)
  Participant 11 - 30 minutes, Day 14: number analyzed (Participants) | 0 | 0 | 1
  Participant 11 - 30 minutes, Day 14 |  |  | 217
  Participant 11 - 60 minutes, Day 14: number analyzed (Participants) | 0 | 0 | 1
  Participant 11 - 60 minutes, Day 14 |  |  | 546
  Participant 11 - 120 minutes, Day 14: number analyzed (Participants) | 0 | 0 | 1
  Participant 11 - 120 minutes, Day 14 |  |  | 1090
  Participant 11 - 180 minutes, Day 14: number analyzed (Participants) | 0 | 0 | 1
  Participant 11 - 180 minutes, Day 14 |  |  | 1610
  Participant 11 - <6 hours (HR) of 2nd dose, Day 14: number analyzed (Participants) | 0 | 0 | 1
  Participant 11 - <6 hours (HR) of 2nd dose, Day 14 |  |  | 670
  Participant 11 - PRE, Day 7: number analyzed (Participants) | 0 | 0 | 1
  Participant 11 - PRE, Day 7 |  |  | 5140
  Participant 11 - 30 minutes, Day 7: number analyzed (Participants) | 0 | 0 | 1
  Participant 11 - 30 minutes, Day 7 |  |  | 7390
  Participant 11 - Cycle 1 Day 1 (C1D1), Treatment held: number analyzed (Participants) | 0 | 0 | 1
  Participant 11 - Cycle 1 Day 1 (C1D1), Treatment held |  |  | 7470
  Participant 11 - End of treatment (EOT): number analyzed (Participants) | 0 | 0 | 1
  Participant 11 - End of treatment (EOT) |  |  | 1.53
  Participant 12 - PRE, Day 14: number analyzed (Participants) | 0 | 0 | 1
  Participant 12 - PRE, Day 14 |  |  | NA — Below quantifiable limit (BQL)
  Participant 12 - 30 minutes, Day 14: number analyzed (Participants) | 0 | 0 | 1
  Participant 12 - 30 minutes, Day 14 |  |  | 54.7
  Participant 12 - 60 minutes, Day 14: number analyzed (Participants) | 0 | 0 | 3
  Participant 12 - 60 minutes, Day 14 |  |  | 104
  Participant 12 - 120 minutes, Day 14: number analyzed (Participants) | 0 | 0 | 1
  Participant 12 - 120 minutes, Day 14 |  |  | 165
  Participant 12 - 180 minutes, Day 14: number analyzed (Participants) | 0 | 0 | 1
  Participant 12 - 180 minutes, Day 14 |  |  | 795
  Participant 12 - <6 hours (HR) of 2nd dose, Day 14: number analyzed (Participants) | 0 | 0 | 1
  Participant 12 - <6 hours (HR) of 2nd dose, Day 14 |  |  | 1380
  Participant 12 - PRE, Day 7: number analyzed (Participants) | 0 | 0 | 1
  Participant 12 - PRE, Day 7 |  |  | 5100
  Participant 12 - 30 minutes, Day 7: number analyzed (Participants) | 0 | 0 | 1
  Participant 12 - 30 minutes, Day 7 |  |  | 4920
  Participant 12 - PRE, Cycle 1 Day 1 (C1D1): number analyzed (Participants) | 0 | 0 | 1
  Participant 12 - PRE, Cycle 1 Day 1 (C1D1) |  |  | 7120
  Participant 12 - End of infusion (EOI), C1D1: number analyzed (Participants) | 0 | 0 | 1
  Participant 12 - End of infusion (EOI), C1D1 |  |  | 6320
  Participant 12 - PRE, C1D15, M7824 held: number analyzed (Participants) | 0 | 0 | 1
  Participant 12 - PRE, C1D15, M7824 held |  |  | 14.6
  Participant 12 - End of treatment (EOT), C2D1: number analyzed (Participants) | 0 | 0 | 1
  Participant 12 - End of treatment (EOT), C2D1 |  |  | 2.13

9. Secondary Outcome: Pharmacodynamic Profile of SX-682 as a Single Agent and in Combination
Description: as for outcome 8
Time Frame: Predose, 30 minutes, 60 minutes, 120 minutes, <6 hours of 2nd dose, and end of infusion (EOI)
Population: No blood samples were collected because the study was closed prior to enrollment of any participants who would have received combination. Early closure was due to a safety stopping rule pre-specified in the protocol. Since no participants received SX-682 treatment in combination, with bintrasfusp alfa and CV-301, PK analysis cannot be performed as outlined in the study objectives. We cannot assess this endpoint without samples from participants treated with SX-682 + bintrasfusp alfa and CV-301.
Arm/Group | Phase I Dose Level 1(DL1) 25mg SX-682 Monotherapy Sequentially Foll/by 1200mg BinTraFusp Alfa +CV301 | Phase I Dose Level 2 (DL2) 50 mg SX-682 Sequentially Followed by 1200mg BinTraFusp Alfa + CV301 | Phase I Dose Level 3 (DL3) 100 mg SX-682 Sequentially Followed by 1200mg BinTraFusp Alfa +CV301
Number analyzed (Participants) | 0 | 0 | 0

10. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 5 months and 9 days, 13 months and 17 days, and 6 months and 1 day for DL1, DL2, and DL3 respectively. Adverse events were assessed beyond the primary completion date.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level 1(DL1) 25mg SX-682 Monotherapy Sequentially Foll/by 1200mg BinTraFusp Alfa +CV301 | Phase I Dose Level 2 (DL2) 50 mg SX-682 Sequentially Followed by 1200mg BinTraFusp Alfa + CV301 | Phase I Dose Level 3 (DL3) 100 mg SX-682 Sequentially Followed by 1200mg BinTraFusp Alfa +CV301
Number analyzed (Participants) | 3 | 6 | 3
Participants | 3 | 6 | 3

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 5 months and 9 days, 13 months and 17 days, and 6 months and 1 day for DL1, DL2, and DL3 respectively. Adverse events were assessed beyond the primary completion date.
Arm/Group | Phase I Dose Level 1(DL1) 25mg SX-682 Monotherapy Sequentially Foll/by 1200mg BinTraFusp Alfa +CV301 | Phase I Dose Level 2 (DL2) 50 mg SX-682 Sequentially Followed by 1200mg BinTraFusp Alfa + CV301 | Phase I Dose Level 3 (DL3) 100 mg SX-682 Sequentially Followed by 1200mg BinTraFusp Alfa +CV301
All-Cause Mortality (participants affected / at risk) | 1/3 | 3/6 | 2/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/6 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dose Level 1(DL1) 25mg SX-682 Monotherapy Sequentially Foll/by 1200mg BinTraFusp Alfa +CV301 (N=3) | Phase I Dose Level 2 (DL2) 50 mg SX-682 Sequentially Followed by 1200mg BinTraFusp Alfa + CV301 (N=6) | Phase I Dose Level 3 (DL3) 100 mg SX-682 Sequentially Followed by 1200mg BinTraFusp Alfa +CV301 (N=3)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Disease progression (General disorders) | 0 (0) | 1 (1) | 0 (0)
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatobiliary disorders - Other, hepatobiliary dilatation (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, COVID-19 infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dose Level 1(DL1) 25mg SX-682 Monotherapy Sequentially Foll/by 1200mg BinTraFusp Alfa +CV301 (N=3) | Phase I Dose Level 2 (DL2) 50 mg SX-682 Sequentially Followed by 1200mg BinTraFusp Alfa + CV301 (N=6) | Phase I Dose Level 3 (DL3) 100 mg SX-682 Sequentially Followed by 1200mg BinTraFusp Alfa +CV301 (N=3)
Abdominal pain (Gastrointestinal disorders) | 1 (3) | 1 (1) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (2) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 3 (4) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
Fatigue (General disorders) | 1 (1) | 4 (4) | 2 (2)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 2 (5) | 2 (5) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, Mucosal bleeding-hematuria (General disorders) | 1 (1) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) | 0 (0) — mucosal bleeding-Epistaxis when blowing nose
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) | 0 (0) — mucosal bleeding-Gingival bleed with brushing teeth
Headache (Nervous system disorders) | 1 (1) | 2 (3) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 2 (6) | 5 (10) | 2 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 1 (2) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Metabolism and nutrition disorders - Other, Increased thirst (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Keratoacanthomas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — Keratoacanthomas? arms, legs, torso
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (3) | 2 (2)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, abnormal urinalysis, bilirubin present (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Sebaceous cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-17): https://cdn.clinicaltrials.gov/large-docs/83/NCT04574583/Prot_SAP_002.pdf
  • Informed Consent Form (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT04574583/ICF_001.pdf